CLINICAL TRIAL: NCT01255644
Title: Treatment of Chronic Lymphocytic Leukemia With the Use of an Antiviral Compound - a Proof of Principle Study
Brief Title: Antiviral Treatment of Chronic Lymphocytic Leukemia
Acronym: VGCV-CLL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Dr. Christoph Steininger, Principal Investigator, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT_2010-021786-78
Record Dates: First submitted 2010-12-06; First posted 2010-12-07 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Valganciclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Antiviral drug (Experimental)
  Interventions: Drug: Valganciclovir

INTERVENTIONS:
Drug: Valganciclovir — 900 mg every 24 hours per os, day 1 through 90
  Other Names: Valcyte

SUMMARY:
Chronic lymphocytic leukemia (CLL) is increasingly believed to be closely related to chronic stimulation of healthy B-cells. Identification of antigen(s) are relevant for the stimulation of CLL precursor cells is therefore of high interest. The investigators found recently evidence that a herpes virus is involved in this process of stimulation. Consequently, elimination of the antigenic stimulation of leukemic cells by this herpes virus may be expected to reduce or even inhibit propagation of leukemic cells. The investigators hypothesize that inhibition of CMV replication by a short course of antiviral treatment may reduce significantly proliferation rates of leukemic cells. To test this hypothesis, the investigators will treat 20 CLL patients with an antiviral drug for 3 months in a proof-of-concept clinical trial and leukemic cell counts measured before and after antiviral treatment. Antiviral treatment has the potential to treat the disease at its origin and therefore more efficiently than conventional chemotherapeutic regimens.

ELIGIBILITY:
Inclusion Criteria:

* CLL confirmed by immunophenotyping and a relative preponderance of leukemic cells of >70%
* ANC >1.500 /µl, Thrombocyte count >100.000 /µl und hemoglobin value >11 g/dl
* CLL patients with expression of immunoglobulin heavy chains (IGHV) 1-69 or 3-21
* Seropositive for CMV-specific IgG-antibodies
* Older than 18 years of age
* Written informed consent
* Able to comply with the protocol
* If female, should not be pregnant or be breast-feeding. Women of child-bearing age must have a negative serum pregnancy test within 28days prior to enrollment into the study, if a serum pregnancy test is not performed within 7 days prior first IMP administration; a confirmatory urine test is required.

Exclusion Criteria:

* Indications for treatment of CLL (advanced stages of the disease)
* Having receiving chemotherapy for CLL within 3 months prior to enrollment
* Having received antiviral drugs or i.v. immunoglobulins within 3 months prior to enrollment
* Significant thrombocytopenia (<100.000/µl) or anemia (Hb < 11 g/dl)
* Women of child bearing age not using effective contraception
* Pregnant of lactating female (as determined by a positive pregnancy test at screening or within 7 days prior to first IMP administration)
* Known hypersensitivity to drug or its excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-12; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Leukocyte count | Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Steininger, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Background] Steininger C, Rassenti LZ, Vanura K, Eigenberger K, Jager U, Kipps TJ, Mannhalter C, Stilgenbauer S, Popow-Kraupp T. Relative seroprevalence of human herpes viruses in patients with chronic lymphocytic leukaemia. Eur J Clin Invest. 2009 Jun;39(6):497-506. doi: 10.1111/j.1365-2362.2009.02131.x. PMID 19490058
- [Background] Vanura K, Le T, Esterbauer H, Spath F, Porpaczy E, Shehata M, Eigenberger K, Hauswirth A, Skrabs C, Kromer E, Schwarzinger I, Streubel B, Steininger C, Fonatsch C, Stilgenbauer S, Wagner O, Gaiger A, Jager U. Autoimmune conditions and chronic infections in chronic lymphocytic leukemia patients at diagnosis are associated with unmutated IgVH genes. Haematologica. 2008 Dec;93(12):1912-6. doi: 10.3324/haematol.12955. Epub 2008 Oct 6. PMID 18838479